CLINICAL TRIAL: NCT01953406
Title: Phase II Study Evaluating the Efficacy of 5-fluorouracil/Mitomycin for the Patients With Pulmonary Metastasis of Hepatocellular Carcinoma Who Had Progressive Disease With Sorafenib
Brief Title: The Efficacy of 5-fluorouracil/Mitomycin for the Patients With Pulmonary Metastasis of Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants were enrolled. Therefore, we stop this study, prematurely.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Hwan Yoon, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUNG M_FM
Record Dates: First submitted 2013-09-21; First posted 2013-10-01 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Hepatocellular Carcinoma; Lung Metastasis
Keywords: hepatocellular carcinoma; lung metastasis; 5-fluorouracil/mitomycin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Fluorouracil; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The 5-fluorouracil/mitomycin group (Experimental): Systemic chemotherapy with 5-fluorouracil/mitomycin 5-fluorouracin 15mg/kg/day D1-6 civ + Mitomycin 4mg/day iv push D1,4 till progression, every 4 weeks
  Interventions: Drug: 5-fluorouracil; Drug: Mitomycin

INTERVENTIONS:
Drug: 5-fluorouracil — 5-fluorouracin 15mg/kg/day D1-6 civ till progression, every 4 weeks
  Other Names: 5-FU
Drug: Mitomycin — Mitomycin 4mg/day iv push D1,4 till progression, every 4 weeks

SUMMARY:
The aim of this study is to evaluate the efficacy of 5-fluorouracil + Mitomycin for the patients with pulmonary metastasis of hepatocellular carcinoma who had progressive disease with sorafenib.

DETAILED DESCRIPTION:
Extrahepatic metastasis of hepatocellular carcinoma has recently been paradoxically increasing due to increased survival with effective locoregional therapies. Sorafenib is the first systemic agent that has demonstrated a significant survival benefit in patients with advanced HCC; however, the modest improvement of 3 months is far from satisfactory. There is no convincing evidence, to date, that systemic chemotherapy when tumor progresses after sorafenib therapy improves overall survival. The combination of anticancer agents is important to achieve favourable clinical results. For patients with metastatic liver cancer or HCC, some studies have discussed the effectiveness of 5-fluorouracil/mitomycin(FM). However, few studies have examined the actual FM regimen for HCC.

The aim of this study is to evaluate the efficacy of 5-fluorouracil/mitomycin for the patients with pulmonary metastasis of hepatocellular carcinoma who had progressive disease with sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received previous local therapy treatments for the intrahepatic hepatocellular carcinoma (RFA, PEI, cryoablation, surgery, resection) and who don't have any viable intrahepatic tumor within 3 months of imaging (dynamic liver CT or liver MRI) after the locoregional therapy
* Patients who have measurable lung metastasis
* Patients who have received their last dose of sorafenib more than 14 days before and who had progressive disease of lung metastasis with sorafenib
* Patients who have risk factors of hepatocellular carcinoma (chronic hepatitis B, chronic hepatitis C, liver cirrhosis)
* Age : 18 years to 80 years
* ECOG Performance Status of 0 to 2
* Child-Pugh class A,B (Child-Pugh score 5-9)
* Adequate bone marrow, liver function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * WBC count > 1,000/mm3
  * Absolute neutrophil count > 500/mm3
  * Hb > 7.0 g/dL
  * Platelet count > 50,000 /mm3
  * Bilirubin < 3 mg/dL
  * Adequate clotting function: INR < 2.3 or < 6sec

Exclusion Criteria:

* Child-Pugh score > 10
* ECOG Performance Status > 3
* History of organ allograft
* Patients with uncontrolled co-morbidity which needs treatment
* Patients who have received prior systemic chemotherapy except sorafenib

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Time-to-progression(TTP)of lung metastasis | every 12 weeks, up to 36 weeks

SECONDARY OUTCOMES:
Overall survival | every 12 weeks, up to 36 weeks
Response rates(CR + PR)of lung metastasis | every 12 weeks, up to 36 weeks
progression free survival | every 12 weeks, up to 36 weeks
Time to recurrence of intrahepatic tumor | every 12 weeks, up to 36 weeks
Disease control rates (CR + PR + SD)of lung metastasis | every 12 weeks, up to 36 weeks

OTHER OUTCOMES:
Adverse Events | every 12 weeks, up to 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hwan Yoon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea